CLINICAL TRIAL: NCT05622747
Title: The Time Course of Cardiovascular Function, Cognitive Function and Heat Shock Proteins in Response to Acute Passive Heating in Older Adults
Brief Title: Acute Passive Heating in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Responsible Party: Principal Investigator, Ant Shepherd, Senior Lecturer in Physical Activity, Exercise and Health, University of Portsmouth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UoPAPHHOA
Record Dates: First submitted 2022-11-08; First posted 2022-11-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-03

CONDITIONS: Aging
Keywords: Passive heating; Endothelial function; Heat shock proteins; Cognitive function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Passive heating intervention (Experimental): 1 h hot water immersion (to the clavicle, @40°C, rectal temperature ~38.5°C and <39°C)
  Interventions: Other: Passive heating

INTERVENTIONS:
Other: Passive heating — 1 h hot water immersion (to the clavicle, @40°C, rectal temperature ~38.5°C and <39°C)

SUMMARY:
Aging is associated with a decline in cardiovascular health, cognitive function and losses in muscle strength, with half or more of those over age 65 suffering from two or more comorbidities (e.g., heart disease, type 2 diabetes). The worldwide population of older adults is growing rapidly, with one in six people expected to be over age 65 by 2050. This will place further financial burden from chronic diseases on already stressed healthcare systems. While studies show that frequent exercise is an effective way for older adults to maintain or improve cardiovascular and metabolic health, older individuals are less physically active and do not adhere well to exercise programs, often due to physical or medical limitations. Therefore, alternative methods for older adults to get the same health benefits as exercise require further exploration. Recent work has shown a single session of passive heat therapy could be an alternative way to improve cardiovascular health and cognitive function in various populations, however, the length of time that these benefits last is yet to be explored.

DETAILED DESCRIPTION:
Aging is associated with declines in cardiovascular health and cognitive function as well as chronic inflammation and the development of neurodegenerative conditions such as Alzheimer's and Parkinson's disease. Additionally, ageing results in a loss of muscle size and strength, commonly referred to as sarcopenia, leading to increased risk of falls or adverse exercise-related events. It is well understood that frequent exercise improves cardiovascular and metabolic health whilst lowering the risk of disease and all-cause mortality, acting as a treatment for many different health conditions. Despite the evidence of its efficacy, many individuals struggle with adherence to exercise programmes, particularly older adults and clinical populations, with many individuals within these populations unable to perform exercise due to physical limitations or medical contraindications. With one in six people expected to be over the age of 65 years by 2050 and corresponding increases in non-communicable diseases (e.g., cancer, diabetes, cardiovascular disease) anticipated from this aging population, the development of adjunct treatments or alternatives to exercise to improve general health in older populations is needed.

Recent work has shown one such potential solution could be the use of passive heat therapy (PHT) (e.g., hot water immersion, sauna), which can achieve health benefits comparable to exercise. Acute PHT induces vascular improvements including increased blood flow, reduced blood pressure. and macro- and microvascular dilator function in various populations. Acute PHT has also been shown to increase reaction time, while mixed results have been seen in its effect on executive function in both young and older populations. The mechanisms for these improvements, however, are currently unclear, and may be related to increases in nitric oxide activity or reductions in biomarkers of inflammation.

One potential mechanism for the physiological benefits obtained from PHT is the increase of cytoprotective heat shock proteins (HSP) (specifically HSP27, HSP60, HSP70 and HSP90) intracellularly (i) and extracellularly (e) in response to increases in deep body temperature. Increases in the expression of these HSPs have been shown to play a role in reducing inflammation and protecting the vasculature via increases in endothelial nitric oxide synthase activity. Increased HSP concentrations may also prevent the accumulation of harmful biomarkers in the brain that play a role in cognitive decline and development of neurodegenerative diseases. There is also evidence that increased preoperative levels of both iHSP70 and eHSP70 are correlated with improved postoperative outcomes following cardiac surgery. Aging, however, is associated with a reduction in HSP transcription activity in various tissues, resulting in an impaired heat shock response and development of a pro-inflammatory state.

Previous work using acute hot water immersion has shown mixed results, with various studies showing increases in eHSP70, iHSP70 and iHSP90, while others have reported no change in expression. Heating stimuli applied in these studies has varied in magnitude, duration and whole body or not, and measurements of HSPs have taken place at various time points before, during and after PHT. Therefore, it is possible that upregulation of HSPs may have been missed, as no time course relationship exists between a single bout of PHT and upregulation of HSPs. Additionally, the duration for acute vascular and cognitive benefits from PHT and when function is returned to baseline is yet to be determined. A time course relationship study to determine the peak HSP response to acute passive heat therapy in older adults would provide insight into the relationship between acute changes in vascular or cognitive function and concurrent upregulation of both intracellular and extracellular HSPs, as well as its potential implications for improved surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 55
* Free from cardiometabolic disease
* Body mass index of 18-35 kg/m2
* Receipt of a normal 12-lead ECG approved by the School Independent Medical Officer
* Capacity to understand and provide their written, informed consent to participate in the study protocol

Exclusion Criteria:

* Unable to understand or cooperate with the study protocol due to learning difficulties or otherwise
* Any current, or past medical (last five years), history of any cardiovascular, respiratory, cancer, renal, hepatic, gastrointestinal, haematological, lymphatic, neurological, psychiatric, or any other disease or diseases.
* Any regular medication for the last five years (not including acute courses of treatment of less than one month for discrete, resolved conditions).
* Medications that may influence physiological responses to the passive heating intervention Uncontrolled hypertension (≥ 150 mmHg systolic and/or ≥ 90 mmHg diastolic)
* Body mass index of > 35 kg/m2
* Recent long-term exposure to a hot climate (within the previous three months)
* Current smoker (or have stopped smoking within the previous three months)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Percentage change in brachial artery diameter and return to baseline as assessed by ultrasound.

SECONDARY OUTCOMES:
Brachial and carotid artery blood flow velocity | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Change from baseline in blood flow velocity of the brachial artery and right common carotid artery as assessed via ultrasound. cm/s is the unit.
Carotid vessel diameter | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Change in vessel diameter of the right common carotid artery and return to baseline as assessed via ultrasound. mm is the unit.
Carotid intima-media thickness | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Change in intima-media thickness of the right common carotid artery and return to baseline as assessed via ultrasound. mm is the unit.
Carotid compliance | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Change in compliance of the right common carotid artery and return to baseline as assessed via ultrasound. µm^2 per kilopascal is the unit.
Carotid distensibility | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Change in distensibility of the right common carotid artery and return to baseline as assessed via ultrasound. 10^-3/kPa is the unit.
Carotid stiffness | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Change in stiffness of the right common carotid artery and return to baseline as assessed via ultrasound. Meters per second is the unit.
Microvascular function | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Change in microvascular function and return to baseline as assessed via iontophoresis on the forearm with acetylcholine (Ach) and Insulin, Area under the curve is the unit.
Stroke volume | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Change in stroke volume and return to baseline measured noninvasively via thoracic impedance. mL/m^2 is the unit
Total peripheral resistance | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Change in total peripheral resistance and return to baseline measured noninvasively via thoracic impedance
Cardiac output | Pre hot water immersion, then 1 hour, 3 hours, 24 hours and 48 hours post
  Change in cardiac output and return to baseline measured noninvasively via thoracic impedance. L/min is the unit.
Intracellular HSP27 concentration | Pre hot water immersion, then immediately post, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours post
  Change in iHSP27 concentration and return to baseline. Measured via immunoblotting in peripheral blood mononuclear cells (PBMCs).
Intracellular HSP60 concentration | Pre hot water immersion, then immediately post, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours post
  Change in iHSP60 concentration and return to baseline. Measured via immunoblotting in peripheral blood mononuclear cells (PBMCs).
Intracellular HSP70 concentration | Pre hot water immersion, then immediately post, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours post
  Change in iHSP70 concentration and return to baseline. Measured via immunoblotting in peripheral blood mononuclear cells (PBMCs).
Intracellular HSP90 concentration | Pre hot water immersion, then immediately post, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours post
  Change in iHSP90 concentration and return to baseline. Measured via immunoblotting in peripheral blood mononuclear cells (PBMCs).
Plasma eHSP27 concentration | Pre hot water immersion, then immediately post, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours post
  Change in plasma eHSP27 concentration and return to baseline. Measured via ELISA.
Plasma eHSP60 concentration | Pre hot water immersion, then immediately post, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours post
  Change in plasma eHSP60 concentration and return to baseline. Measured via ELISA.
Plasma eHSP70 concentration | Pre hot water immersion, then immediately post, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours post
  Change in plasma eHSP70 concentration and return to baseline. Measured via ELISA.
Plasma eHSP90 concentration | Pre hot water immersion, then immediately post, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours post
  Change in plasma eHSP90 concentration and return to baseline. Measured via ELISA.
Reaction time | Pre hot water immersion, then immediately post, 3 hours, 24 hours and 48 hours post
  Change in reaction time and return to baseline as assessed using ANAM: Automated Neurophysiological Assessment Metrics.
Logical reasoning | Pre hot water immersion, then immediately post, 3 hours, 24 hours and 48 hours post
  Change in logical reasoning and return to baseline as assessed using ANAM: Automated Neurophysiological Assessment Metrics.
Memory | Pre hot water immersion, then immediately post, 3 hours, 24 hours and 48 hours post
  Change in memory function and return to baseline as assessed using ANAM: Automated Neurophysiological Assessment Metrics.
Cerebral oxygenation | Pre hot water immersion, then immediately post, 3 hours, 24 hours and 48 hours post
  Change in cerebral oxygenation and return to baseline. Assessed using Near-infrared spectroscopy (NIRS) attached to the forehead

CONTACTS AND LOCATIONS:
Locations (1):
- Spinnaker Building, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All data will be anonymized and raw data uploaded to the University of Portsmouth repository.
Supporting Information: Study Protocol
Time Frame: After data has been collected and analyzed it will be available indefinitely.
Access Criteria: Available to public at repository website